CLINICAL TRIAL: NCT00581724
Title: Pain in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Beth Israel Medical Center (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 07-068
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer; Colorectal Cancer; Prostate Cancer; Head and Neck Cancer; Lung Cancer
Keywords: breast cancer; Colorectal cancer; Prostate cancer; Head and Neck cancer; Lung cancer; cancer survivors; 07-068; quality of life; Pain in cancer survivors
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Head and Neck Neoplasms; Lung Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: First 50 breast cancer survivors and then after demonstrating feasibility of the study design in the first 50 participants, recruitment will be opened to the other services Colorectal, Genitourinary, Head and Neck, and Thoracic.
  Participants will be recruited in allotments of 50 patients from each service.
  Interventions: Behavioral: Telephone interview or self report survey.

INTERVENTIONS:
Behavioral: Telephone interview or self report survey. — We estimate that the completion time for the telephone interview or self-report survey will be 45-60 minutes.

SUMMARY:
The purpose of this study is to find out about the pain and quality of life of individuals who are adult cancer survivors. By quality of life, we mean how you are feeling about different aspects of your life, including your physical health, your emotional health, and your ability to carry out daily activities. We are interested in people's opinions about their quality of life, as well as the factors that affect their quality of life. In addition, learning about pain will help us to develop new services for adult cancer survivors.

DETAILED DESCRIPTION:
The main objective of the proposed study is to identify the prevalence of persistent pain in a sample of adult cancer survivors. Currently, there is a lack of comprehensive information about pain in the cancer survivor population. Although prior studies have assessed pain syndromes in breast and lung cancer survivors (e.g., post-mastectomy and post-thoracotomy pain), there is a lack of information about the prevalence and characteristics of post-treatment pain in other subpopulations of survivors. To address this knowledge gap, a random sample of cancer survivors who are from 1 to 10 years post-treatment completion and who were treated at Memorial Sloan-Kettering Cancer Center will complete a telephone-administered pain interview and assessment battery focusing on pain, quality of life, and psychological distress. Our initial recruitment and evaluation will begin in 50 breast cancer survivors and then will expand 50 survivors in each of the other services Colorectal, Genitourinary, Head and Neck, and Thoracic in allotments of 50 participants each. We estimate that the completion time for the interview and assessment battery will range from 45 to 60 minutes. This telephone-based survey will identify vulnerable subgroups of patients with persistent pain and provide a knowledge base for future research on the prevalence and risk factors for post-treatment pain in the cancer survivor population.

ELIGIBILITY:
Inclusion Criteria:

* Cancer treatment at MSKCC
* Are from 1 to 10 years post-treatment completion at the time of study recruitment
* No evidence of disease (NED) at the time of assessment;
* Over 18 years of age
* Can be reached by telephone
* Able to provide informed consent
* Able to speak and read English
* Cancer survivors who received adjuvant therapies outside MSKCC will be asked to self-report the type and duration of cancer treatments received.

Exclusion Criteria:

* Undergoing active cancer treatment (ongoing tamoxifen use, hormone replacement therapy or use of biologics are permitted)
* Evidence of encephalopathy, psychotic illness or cognitive impairment severe enough to preclude giving informed consent to the study staff, or completing the survey instruments of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer survivors that were treated for cancer at Memorial Sloan-Kettering Cancer Center (MSKCC) and it has been at least a year since you completed treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Descriptive statistics will be generated to describe the prevalence of pain and its psychosocial correlates. | 1 to 10 years post-treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Steven Passik, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States